CLINICAL TRIAL: NCT01451840
Title: Efficacy of Alkalinized Lidocaine in the Endotracheal Tube Cuff Compared to a Bolus Dose of Intravenous Remifentanil on the Incidence of Coughing During Emergence of Anesthesia
Brief Title: Efficacy of Alkalinized Lidocaine Compared to Remifentanil on the Incidence of Coughing During Emergence of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NM2012-001
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Cough; Anesthesia
MeSH Terms: conditions — Cough | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil 0.25 mcg/kg (Active Comparator): Administration of a bolus dose of intravenous remifentanil before emergence of a desflurane-based anesthesia
  Interventions: Drug: Remifentanil
- Alkalinized lidocaine (Experimental): Administration of alkalinized lidocaine in the endotracheal tube cuff
  Interventions: Drug: Alkalinized lidocaine

INTERVENTIONS:
Drug: Remifentanil — Bolus dose of intravenous remifentanil 0.25 mcg/kg given once before emergence of general anesthesia
  Arms: Remifentanil 0.25 mcg/kg
Drug: Alkalinized lidocaine — Administration of alkalinized lidocaine in the endotracheal tube cuff
  Arms: Alkalinized lidocaine

SUMMARY:
This study is designed to compare the effects of alkalinized lidocaine in the endotracheal tube cuff to a bolus dose of remifentanil given prior to the emergence of anesthesia:

* on the incidence of perioperative coughing
* on the time needed for the emergence of a desflurane-based anesthesia
* on the incidence of sore throat after extubation.

The investigators hypothesis is that the use of alkalinized lidocaine in the endotracheal tube cuff will reduce the incidence of perioperative coughing after a desflurane-based anesthesia.

DETAILED DESCRIPTION:
Emergence is an important period of general anesthesia during which several problems can occur. Coughing, hypertension, tachycardia and agitation have been observed during emergence of general anesthesia.

Desflurane is a newer volatile agent allowing early recovery from anesthesia. This agent has led to earlier discharge and more rapid resumption of normal activities after surgery. However, an incidence of coughing around 70% has been reported after a desflurane-based anesthesia. Different techniques and drugs have been studied to reduce coughing during emergence.

Among others, the role of lidocaine given intravenously, topically, or intracuff has been studied. The use of intracuff alkalinized lidocaine has been proven effective to reduce the incidence of coughing during emergence of anesthesia.

Furthermore, there is some evidence supporting the administration of intravenous opioids prior to emergence of general anesthesia to reduce perioperative coughing, agitation and hemodynamic stimulation. However, depending on the type of opioids given, this may delay the emergence from anesthesia. The effect of a remifentanil infusion given in combination with isoflurane as the volatile agent has been shown to reduce the incidence of perioperative coughing without delaying the emergence of anesthesia. Bolus doses of remifentanil have also been proven effective to reduce the hemodynamic response to extubation.

The effect of these two modalities (alkalinized lidocaine and remifentanil) have never been compared. This study will assess their efficacy to prevent perioperative coughing after a desflurane-based anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Physical status 1-3
* Patients undergoing elective surgery under general anesthesia requiring oral endotracheal intubation (excluding head and neck surgery)
* Expected duration of surgery of at least 1.5 hour.

Exclusion Criteria:

* Current use of ACE inhibitor
* Chronic cough
* Asthma or severe pulmonary disease
* Pulmonary tract infection
* Anticipated difficult intubation
* Current use of opioids
* Current use of cough medicine
* Contraindication to remifentanil, lidocaine
* Pregnancy
* Symptomatic cardiac, renal or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing during emergence and after extubation | From emergence until 10 minutes after extubation

SECONDARY OUTCOMES:
Time to emergence | From the discontinuation of Desflurane until extubation
Incidence of sore throat one hour after extubation | Assessed one hour after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD,FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada